CLINICAL TRIAL: NCT03517917
Title: Prospective Collection of Donor Tissue and Whole Blood or Leukapheresis Product From Patients With Solid Tumours to Enable Development of Methods for the Manufacturing of Clonal Neoantigen T Cell Products (cNeT)
Brief Title: Prospective Tissue Collection Research Protocol
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: ATX-MAP-001
Record Dates: First submitted 2018-04-25; First posted 2018-05-08 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Solid Tumor

GROUPS / COHORTS (1):
- Arm 1: Tumour tissue, blood and leukapheresis collection to enable a manufacturing process for immunotherapies to be developed.
  Interventions: Other: Tumour tissue collection

INTERVENTIONS:
Other: Tumour tissue collection — Collection of tumour tissue and blood

SUMMARY:
This is a multi-solid tumour research study which collects tumour samples from patients alongside a matched whole blood, and/or leukapheresis product for the development of manufacturing processes for potential immunotherapies.

DETAILED DESCRIPTION:
During standard of care surgery tumour samples which are surplus to the requirements of the patients diagnostic/treatment pathway will be procured along with a matched whole blood and/or leukapheresis sample. In some instances patients may consent to provide a non-standard of care, non-invasive research biopsy.

Within 28-42 days following procurement of samples patients will be required to participate in a safety follow up call for assessment of any procedure related adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Written informed patient consent for tissue, blood collection or leukapheresis, including storage and manipulation.
* Suspected or confirmed diagnosis of selective solid tumours with either primary, recurrent or metastatic disease.
* Patient is scheduled for surgical excision and/or collection of multiple tissue samples via image or device guided biopsy, has a superficial skin or subcutaneous lymph node metastasis that can be safely accessed for the purposes of the study.
* Haemoglobin(Hb) ≥ 10g/dL without transfusion support for at least 3 weeks (for patients donating whole blood).

White cell count ≥ 3 x 10^9/L (for patients donating whole blood).

* For selected solid tumours and leukapheresis procedure additional inclusion criteria apply.

Exclusion Criteria:

* Clinical status precludes surgical removal of, or collection of multiple biopsies from, accessible tumour tissue.
* Inadequate peripheral venous access precluding collection of blood.
* Pregnant or breastfeeding women.
* Known/laboratory confirmed diagnosis of an active infectious disease to include Hepatitis B and C, human immunodeficiency virus infection (HIV1/2), Human t-lymphotropic virus (HTLV I/II) and syphilis.
* Patients who are currently participating in a clinical trial involving an unlicensed medical product.
* Patients who have received any cytotoxic therapy (including investigational products) within three weeks prior to tissue procurement.
* Patients receiving immunosuppressive treatments or who require regular treatment with steroids at a dose higher than prednisolone 10 mg/day (or equivalent).
* Any medical reason why, in the opinion of the investigator, the patient should not participate in this study.
* For selected solid tumours and leukapheresis procedure additional exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with solid tumour scheduled for either biopsy or resection of their tumour(s) as part of their standard of care, and patients with superficial skin or subcutaneous lymph node metastasis that can be safely accessed for the purposes of the study.
Sampling Method: Non-Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
Obtaining samples for research | 5 years
  This protocol does not have an analysis primary outcome measure. It will be conducted in accordance with the principles of Good Clinical Practice (GCP), solely for the purpose of obtaining samples for research.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (3):
  - Research Site, New York, New York
  - Research Site, Durham, North Carolina
  - Research Site, Georgetown, Washington
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Madrid
- United Kingdom (7):
  - Research Site, Glasgow
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne
  - Research Site, Southampton
  - Research Site, Uxbridge

REFERENCES:
- See also: Privacy Data — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ATX-MAP-001&attachmentIdentifier=eb3f4be2-9189-4034-bda9-b8f959d2f2f0&fileName=Notification_of_Sponsor_Change_to_Study_Participants_in_the_MAP_Study_(ATX-MAP-001).pdf&versionIdentifier=